CLINICAL TRIAL: NCT05090904
Title: A Phase 2a, Single-Blind, Placebo-Controlled, Parallel-Group Study to Assess Safety, Tolerability, and Pharmacokinetics of Brensocatib Tablets in Adults With Cystic Fibrosis
Brief Title: A Study to Assess the Safety, Tolerability, and Pharmacokinetics of Brensocatib Tablets in Adults With Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INS1007-211
Record Dates: First submitted 2021-10-14; First posted 2021-10-25 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Brensocatib
MeSH Terms: conditions — Cystic Fibrosis | interventions — brensocatib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Brensocatib 10 mg (Experimental): Participants will be administered brensocatib at a dose of 10 mg once per day for 28 days. The participants will be stratified based on cystic fibrosis transmembrane conductance regulators (CFTRs) modulator treatment.
  Interventions: Drug: Brensocatib
- Brensocatib 25 mg (Experimental): Participants will be administered brensocatib at a dose of 25 mg once per day for 28 days. The participants will be stratified based on CFTRs modulator treatment.
  Interventions: Drug: Brensocatib
- Brensocatib 40 mg (Experimental): Participants will be administered brensocatib at a dose of 40 mg once per day for 28 days. The participants will be stratified based on CFTRs modulator treatment.
  Interventions: Drug: Brensocatib
- Brensocatib 65 mg (Experimental): Following review of safety and pharmacokinetic data by the safety review committee, an additional cohort of participants may be administered brensocatib at a dose of 65 mg once per day for 28 days. The participants will be stratified based on CFTRs modulator treatment.
  Interventions: Drug: Brensocatib
- Placebo (Placebo Comparator): Participants will be administered a placebo matching brensocatib once per day for 28 days. The participants will be stratified based on CFTRs modulator treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Brensocatib — Oral tablet
  Other Names: INS1007
  Arms: Brensocatib 10 mg; Brensocatib 25 mg; Brensocatib 40 mg; Brensocatib 65 mg
Drug: Placebo — Oral tablet
  Arms: Placebo

SUMMARY:
The main objective of the study is to evaluate the pharmacokinetics of brensocatib in participants with cystic fibrosis following once daily oral administration of study drug and to evaluate the safety of brensocatib compared to placebo in participants with cystic fibrosis (CF) over the 4-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ≥18 years of age at the time of signing the informed consent.
* Male or female participants with a confirmed diagnosis of CF related lung disease:

  1. Percent predicted forced expiratory volume in 1 second (ppFEV1) between 40% to 90% (inclusive) at Screening Visit and at Baseline.
  2. Stable CF treatment for at least 30 days before screening and willing to remain on a stable regimen throughout the treatment period.
* Has a body mass index ≥18 kg/m^2.
* Male and female participants must use contraceptives that are consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

  1. Male participants, who are not sterile, with female partners of childbearing potential must be using effective contraception from Day 1 to at least 90 days after the last dose.
  2. Women must be postmenopausal (defined as no menses for 12 months without an alternative medical cause), surgically sterile, or using highly effective contraception methods (i.e., methods that alone or in combination achieve <1% unintended pregnancy rates per year when used consistently and correctly) from Day 1 to at least 90 days after the last dose.
* Female participants of childbearing potential must have a negative serum pregnancy test at Screening.
* Male participants with pregnant or nonpregnant women of childbearing potential partners must use a condom.

Exclusion Criteria:

* Severe or unstable CF, per Investigator's judgement.
* Currently being treated for allergic bronchopulmonary aspergillosis or nontuberculous mycobacteria or tuberculosis.
* Active and current infection by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
* History of malignancy in the past 5 years, except completely treated in situ carcinoma of the cervix and completely treated non-metastatic squamous or basal cell carcinoma of the skin.
* Established diagnosis of hepatitis B viral infection or positive for hepatitis B surface antigen (HBsAg) at Screening.
* Established diagnosis of hepatitis C virus (HCV) infection at Screening. Participants positive for hepatitis C antibody are eligible only if HCV RNA is negative.
* History of human immunodeficiency virus (HIV) infection.
* Acute upper or lower respiratory tract infection, pulmonary exacerbation, or changes in therapy (including intravenous and oral antibiotics) for pulmonary disease within 4 weeks prior to Day 1 (administration of the first dose of study drug). Participants meeting this criterion could be rescreened 4 weeks after resolution of symptoms.
* History of prolonged QT/QTc interval with QTcF >480 millisecond (msec) at Screening.
* History of solid organ or hematological transplantation.
* Have diagnosed periodontal disease and are either:

  1. Currently treated by a dentist for this condition or
  2. Expected to have periodontal disease-related procedures within the study period.
* Received any live attenuated vaccine within 4 weeks prior Screening.
* Ongoing participation in another therapeutic clinical study or prior participation in an investigational drug study within 90 days prior to Screening.
* Known history of hypersensitivity to brensocatib or any of its excipients.
* Use of any immunomodulatory agents within 4 weeks before the Screening Visit is prohibited during the study through end of study (including, but not limited to: bortezomib, ixazomib, thalidomide, cyclophosphamide, mycophenolate, Janus kinase inhibitors, interferon gamma (IFN-γ], and azathioprine).
* Continuous use of high-dose non-steroidal anti-inflammatory drugs (NSAIDs) is prohibited during the study through end of study.
* History of alcohol, medication, or illicit drug abuse.
* Current smoker, as defined by Centers for Disease Control and Prevention: An adult who has smoked 100 cigarettes in his or her lifetime and who currently smokes cigarettes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of Brensocatib | Day 1: Predose and 0.5, 1, 2, 4, 6, 8, and 24 hours postdose; Day 28: Predose and at 0.5, 1, 2, 4, 6, 8, 24 and 168 hours postdose
Time to Maximum Plasma Concentration (tmax) of Brensocatib | Day 1: Predose and 0.5, 1, 2, 4, 6, 8, and 24 hours postdose; Day 28: Predose and at 0.5, 1, 2, 4, 6, 8, 24 and 168 hours postdose
Area Under the Concentration-time Curve from Time 0 to 24 Hours Post-dose (AUC0-24) of Brensocatib | Day 1: Predose and 0.5, 1, 2, 4, 6, 8, and 24 hours postdose; Day 28: Predose and at 0.5, 1, 2, 4, 6, 8, 24 hours postdose
Elimination Half-life (t1/2) of Brensocatib | Day 1: Predose and 0.5, 1, 2, 4, 6, 8, and 24 hours postdose; Day 28: Predose and at 0.5, 1, 2, 4, 6, 8, 24 and 168 hours postdose
Number of Participants Who Experience a Treatment-emergent Adverse Event (TEAE) | Day 1 to Day 56

SECONDARY OUTCOMES:
Dose-normalized Maximum Plasma Concentration (Cmax) of Brensocatib | Day 1: Predose and 0.5, 1, 2, 4, 6, 8, and 24 hours postdose; Day 28: Predose and at 0.5, 1, 2, 4, 6, 8, 24 and 168 hours postdose
Dose-normalized Area Under the Concentration-time Curve from Time 0 to 24 Hours Post-dose (AUC0-24) of Brensocatib | Day 1: Predose and 0.5, 1, 2, 4, 6, 8, and 24 hours postdose; Day 28: Predose and at 0.5, 1, 2, 4, 6, 8, 24 hours postdose
Dose-normalized Area Under the Concentration-time Curve from Time 0 to the Time of Last Measurable Concentration (AUClast) of Brensocatib | Day 1: Predose and 0.5, 1, 2, 4, 6, 8, and 24 hours postdose; Day 28: Predose and at 0.5, 1, 2, 4, 6, 8, 24 and 168 hours postdose

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - USA001, Gainesville, Florida
  - USA016, Augusta, Georgia
  - USA025, Glenview, Illinois
  - USA011, Boston, Massachusetts
  - USA023, Ann Arbor, Michigan
  - USA002, St Louis, Missouri
  - USA022, New York, New York
  - USA008, Cleveland, Ohio
  - USA006, Cleveland, Ohio
  - USA018, Portland, Oregon
  - USA009, Charleston, South Carolina
  - USA017, Nashville, Tennessee
  - USA004, Dallas, Texas
  - USA003, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Konstan MW, Tolle JJ, DiMango E, Flume PA, Usansky H, Teper A, Ramirez CN, Flarakos J, Basso J, Li S, Vergara M. A Phase IIa, Single-Blind, Placebo-Controlled, Parallel-Group Study to Assess Safety, Tolerability, and Pharmacokinetics/Pharmacodynamics of Brensocatib in Adults with Cystic Fibrosis. Clin Pharmacokinet. 2025 Oct;64(10):1561-1574. doi: 10.1007/s40262-025-01550-z. Epub 2025 Aug 3. PMID 40753522